CLINICAL TRIAL: NCT03359772
Title: Effectiveness of Balance Training With Kinesthetic Ability Trainer-KAT2000 in Patients With Peripheral Neuropathic Pain: a Randomized Controlled Study
Brief Title: Kinesthetic Ability Trainer for Peripheral Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, ASLIHAN UZUNKULAOGLU, Ufuk University, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30112015-4
Record Dates: First submitted 2017-10-25; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain; Balance; Kinesthetic Ability Trainer; Quality of Life
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): Exercise Only Group
- Group 2 (Active Comparator): Kinesthetic Ability Trainer Group
  Interventions: Other: Kinesthetic Ability Trainer

INTERVENTIONS:
Other: Kinesthetic Ability Trainer — Kinesthetic Ability Trainer
  Arms: Group 2

SUMMARY:
Objective: To determine the effectiveness of balance training with Kinesthetic Ability Trainer 2000 (KAT 2000) in patients with peripheral neuropathic pain related balance disorder.

Methods: A total of 60 patients who developed peripheral neuropathic pain-related balance impairment in the chronic phase due to lumber disc herniation, lumber spondylosis and gonarthrosis were included into this randomized controlled prospective study and randomized into either balance exercises groups or KAT 2000 exercises groups. Balance exercises were given all patients in Group 1 (n=30). In addition to balance exercises, KAT 2000 balance exercises were given all patients in group 2 (n=30). All patients received 45-min individualized training session for three times a week for 4 weeks. Patients were evaluated according to pain, static and dynamic balance and quality of life (QoL).

DETAILED DESCRIPTION:
Neuropathic pain was determined by the Douleur Neuropathique 4 (DN4) questionnaire. Pain severity was assessed by using a visual analogue scale (VAS). KAT 2000 was used to evaluate static and dynamic balance. Dynamic balance and mobility also was assessed using the Berg Balance Scale (BBS) and Time Up and Go (TUG) test. QoL was assessed by using Nottingham Health Profile (NHP). Patients were evaluated at baseline and the end of the 4-week exercise program.

ELIGIBILITY:
Inclusion Criteria:

* DN4 scores ≥4 and moderately impaired balance with a score of 21-40 points on the Berg Balance Scale.

Exclusion Criteria:

* Who had history of previous cerebrovascular events; other neurological, musculoskeletal, inner ear or eye disease that may lead to impaired vision or standing balance.

Ages: 64 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Douleur Neuropathique 4 | 1 months
  Neuropathic pain questionnaire, if Douleur Neuropathique 4 value is 4 of more, there is neuropathic pain

SECONDARY OUTCOMES:
visual analogue scale | 1 months
  for pain evaluation
Berg Balance Scale | 1 months
  for balance evaluation
Time Up and Go Test | 1 months
  for functional evaluation
Nottingham Health Profile | 1 months
  for evaluation of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: DUYGU KERİM, Study Chair — Ufuk University; Saime AY, Study Chair — Ufuk University
Locations (1):
- Ufuk University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No